CLINICAL TRIAL: NCT04025866
Title: The Addition of Aerobic Training to Conventional Rehabilitation After Proximal Femur Fracture: a Randomized Controlled Trial
Brief Title: Addition of Aerobic Training to Conventional Rehabilitation After Femur Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2264 CE
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Intertrochanteric Fractures
Keywords: conventional rehabilitation; arm ergometer; aerobic exercise; intertrochanteric fractures
MeSH Terms: conditions — Hip Fractures | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional rehabilitation (Active Comparator): Conventional rehabilitation treatment for inpatients with femur fracture
  Interventions: Other: Conventional rehabilitation
- Aerobic exercise (Active Comparator): Addition of cycle ergometer for upper limb to conventional rehabilitation treatment for femur fracture
  Interventions: Other: Conventional rehabilitation; Other: Aerobic exercise

INTERVENTIONS:
Other: Conventional rehabilitation — 1h/day for 5 days/week of conventional rehabilitation for femur fracture
Other: Aerobic exercise — 30 min/day of aerobic exercise with arm cycle ergometer added to 1h/day for 5 days/week of conventional rehabilitation for femur fracture
  Arms: Aerobic exercise

SUMMARY:
The primary purpose of this study is to assess the feasibility of an arm cycle ergometer training in subjects with proximal femur fracture surgically treated. The secondary purpose of this randomized controlled clinical trial is to verify whether the addition of aerobic activity can increase motor performance compared to a conventional exercise program in which no aerobic activity is foreseen.

DETAILED DESCRIPTION:
Every year in Italy more than 100,000 persons aged > 65 incur in a hip fracture. The direct costs sustained by National Health System both for hospitalization and rehabilitation following hip fracture in elderly people were estimated in more than one billion euro. Despite incidence rate is decreasing in the last years, the number of hospitalizations for hip fractures is still increasing due to the population aging. Some estimates assume that the number of fractures per year will double by 2050. Observational studies suggest that following hip fracture, only 40-60% of people who survive are likely to reach their prefracture level of mobility. Up to 70% may recover their level of independence for basic activities of daily living and less than half of all people experiencing hip fracture may regain their ability to perform instrumental ADLs.

In Italy, as in Western nations, approximately 10-20% of patients are institutionalized after a hip fracture, which imposes a large cost burden on society.Then, it is widely recognised that a vicious cycle can occur after a hip fracture where pain and hospitalization result in disuse atrophy of muscles and general low level of aerobic fitness which increases the risk of immobility and new fractures. The aerobic fitness level of older adults is a primary determinant of health and morbidity and thus serves as a powerful predictor of quality of life and independent living. Moreover, a number of guidelines recommend that older people, aged over 65, perform at least 150 minutes per week of medium-intensity aerobic activity (where aerobic activity refers to different activities, such as example: walking, cycling, etc.). Elderly subjects undergoing rehabilitation should be physically active to the extent granted by disability and health status.

Contrary to this, patients post-surgery of femur fracture perform low levels of physical activity. In fact patients spend at least 98% of the day during the rehabilitation period in a sitting or lying down position in the bed. On average, these patients take 36 steps a day, which results in less than the 2,000-9,000 steps needed to stay healthy. Indeed deconditioning can be consider a major determining factor for the unsatisfactory recovery of motor skills for patients undergoing femoral surgery during rehabilitation.

There is irrefutable evidence showing the beneficial effects of exercise in both prevention and treatment of several diseases. A lot of studies have shown that both men and women who report increased levels of physical activity and fitness have reductions in relative risk of death (by about 20%-35%). The benefits of exercise are evident, not only in healthy persons but also in patients.

Unfortunately, it is hardly conceivable that these patients could reach, in a hospitalization regime, activity levels equal to those recommended by the guidelines. For all these reasons, the investigators have introduced aerobic training performed with an arm cycle ergometer, in patients hospitalized and subjected to conventional rehabilitation.

The primary purpose of this randomized controlled clinical trial is to verify the feasibility of an aerobic exercise program in subjects with recent proximal femur fracture treated surgically.

The secondary purpose is to verify whether the addition of aerobic activity can increase motor performance compared to a program in which no aerobic activity is foreseen. In particular, the investigators expect the patients belonging to the intervention group to walk faster than those who have performed only conventional physiotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Older men or women aged 65 years and older (with no upper age limit).
2. An intertrochanteric fracture, AO Type 31-A (Muller Classification), confirmed with hip radiographs, surgically repaired by internal fixation.
3. Low energy fracture (defined as a fall from standing height).
4. No other major trauma.
5. Admission to the rehabilitation clinic from 8 to 12 days after the surgery
6. Patients autonomous prior to fracture.
7. Provision of informed consent by patient.

Exclusion Criteria:

1. Associated major injuries of the lower extremity (i.e., ipsilateral and/or contralateral fractures of the foot, ankle, tibia, fibula, or knee; dislocations of the ankle, knee, or hip) or upper extremity (i.e., radius, ulna or humerus fracture).
2. Orthopedic contraindications to mobilization and to lower extremity operated load;
3. Patients with disorders of bone metabolism other than osteoporosis (i.e., Paget's disease, renal osteodystrophy, or osteomalacia).
4. Patients with neurological diseases.
5. Patients with important cardiac diseases.
6. Patients with a pathologic fracture.
7. Patients with subtrochanteric fracture or with a fracture AO Type 31-B or 31-C (Muller Classification).
8. Patients with a previous history of frank dementia.
9. Terminally-ill (life expectation < 6 months).
10. Patients who lived in an institution before the fracture event or were not self-sufficient.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2022-01-11 (Actual)

PRIMARY OUTCOMES:
Analysis of feasibility | Up to 4 weeks
  To assess the feasibility, it will be evaluated:
  1. The eligibility rate (the total number of patients admitted with femur fractures and screening divided by the total number of patients meeting the criteria).
  2. The recruitment rate (the number of patients recruited among those eligible).
  3. The subjects' compliance level will be analyzed dichotomously (no compliance <10 sessions, yes compliance ≥ 10 sessions).
  4. Rate of patients who lost the evaluation at the end of the treatment and at the follow-up after 100 days.
  5. Any negative effects will be recorded and counted. The following types of adverse events will be calculated separately: a) adverse reactions, adverse events, serious adverse events and suspected serious adverse events.
  6. Adherence to treatment: the number of sessions in which patients have reached goal 1) of 30 minutes and 2) intensity between 50%-85% HRmax.

SECONDARY OUTCOMES:
Timed Up and Go (TUG) test | Up to 4 weeks
  TUG is a physical functional measure in which subjects are asked to stand up from a chair, walk 3 m to a horizontal line marked with tape on the floor, turn around, walk back and sit down at a comfortable pace (Podsiadlo et al., 1991).
10-meter Walking Test (10mWT) | Up to 4 weeks
  In the 10mWT the time taken by the patient to travel a linear distance of 10 meters will be timed. During the execution of the test the number of supports will also be recorded, so as to secondly calculate the walking speed (speed (m / s) = space (m) / time (s)), the step length (step length (cm) = 1000 / number of steps) and cadence (cadence (steps / min) = number of steps / time (s) * 60) (Hollman et al., 2008).
Cumulated Ambulation Score - Italian version (CAS-I) | Up to 4 weeks
  The CAS-I is a 3-item scale assessing activities that characterize the patient's basic mobility skills: 1) getting in and out of bed, 2) sit-to-stand from a chair with armrests and 3) walking indoors with the use of appropriate walking aids. Each activity is assessed on a three-point ordinal scale from 0-2 (0 = Not able to, despite human assistance and verbal cueing, 1 = Able to, with human assistance and/or verbal cueing from one or more persons, 2 = Able to safely, without human assistance or verbal cueing, use of a walking aid allowed) resulting in a total daily CAS score ranging from zero to six. The CAS scale showed to be a potentially valuable score for early prediction of short-term postoperative outcome after hip fracture surgery.
Activities-Specific Balance Confidence Scale - 5 levels (ABC 5-levels) | Up to 4 weeks
  The scale led to assessing the confidence of self-reported balance during daily life activities. Each of the 16 items is assigned a score between 0 (no security) and 4 (total security).
Maximum isometric force of the knee extensors | Up to 4 weeks
  The maximum isometric force of the knee extensors will be evaluated pre- and post-training with the use of a manual dynamometer (Roy and Doherty, 2004). The patient will be required to perform a sub-maximal contraction in knee extension, followed by four maximal contractions during which the patient is verbally encouraged by the therapist. The evaluation will be performed first on the healthy limb, then on the operated limb, with a 30-second pause between one contraction and the next. The best value of the 4 tests will then be recorded.
Verbal Ranking Scale (VRS) | Up to 4 weeks
  Pain related to femoral fracture will be assessed using the Verbal Ranking Scale (VRS). Divided over 5 levels (VRS 0-4: 0 = no pain; 1 = mild; 2 = moderate; 3 = strong; 4 = extreme), it allows to record the maximum pain experienced by the patient in the previous 48 hours in the execution of some functional activities, such as sitting, keeping standing and walking (Leino et al., 2011).

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Corna, MD, Principal Investigator — Istituti Clinici Scientifici Maugeri
Locations (1):
- Istituti Clinici Scientifici Maugeri, Veruno, Novara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Piscitelli P, Gimigliano F, Gatto S, Marinelli A, Gimigliano A, Marinelli P, Chitano G, Greco M, Di Paola L, Sbenaglia E, Benvenuto M, Muratore M, Quarta E, Calcagnile F, Coli G, Borgia O, Forcina B, Fitto F, Giordano A, Distante A, Rossini M, Angeli A, Migliore A, Guglielmi G, Guida G, Brandi ML, Gimigliano R, Iolascon G. Hip fractures in Italy: 2000-2005 extension study. Osteoporos Int. 2010 Aug;21(8):1323-30. doi: 10.1007/s00198-009-1084-x. Epub 2009 Oct 7. PMID 19809775
- [Background] Tarantino U, Piscitelli P, Feola M, Neglia C, Rao C, Gimigliano F, Iolascon G. Decreasing trend of hip fractures incidence in Italy between 2007 and 2014: epidemiological changes due to population aging. Arch Osteoporos. 2018 Mar 9;13(1):23. doi: 10.1007/s11657-018-0423-y. PMID 29523987
- [Background] Rossini M, Piscitelli P, Fitto F, Camboa P, Angeli A, Guida G, Adami S. [Incidence and socioeconomic burden of hip fractures in Italy]. Reumatismo. 2005 Apr-Jun;57(2):97-102. doi: 10.4081/reumatismo.2005.97. Italian. PMID 15983632
- [Background] Shah MR, Aharonoff GB, Wolinsky P, Zuckerman JD, Koval KJ. Outcome after hip fracture in individuals ninety years of age and older. J Orthop Trauma. 2001 Jan;15(1):34-9. doi: 10.1097/00005131-200101000-00007. PMID 11147685
- [Background] Magaziner J, Hawkes W, Hebel JR, Zimmerman SI, Fox KM, Dolan M, Felsenthal G, Kenzora J. Recovery from hip fracture in eight areas of function. J Gerontol A Biol Sci Med Sci. 2000 Sep;55(9):M498-507. doi: 10.1093/gerona/55.9.m498. PMID 10995047
- [Background] Norton R, Butler M, Robinson E, Lee-Joe T, Campbell AJ. Declines in physical functioning attributable to hip fracture among older people: a follow-up study of case-control participants. Disabil Rehabil. 2000 May 20;22(8):345-51. doi: 10.1080/096382800296584. PMID 10896094
- [Background] Beaupre LA, Cinats JG, Jones CA, Scharfenberger AV, William C Johnston D, Senthilselvan A, Saunders LD. Does functional recovery in elderly hip fracture patients differ between patients admitted from long-term care and the community? J Gerontol A Biol Sci Med Sci. 2007 Oct;62(10):1127-33. doi: 10.1093/gerona/62.10.1127. PMID 17921426
- [Background] Vergara I, Vrotsou K, Orive M, Gonzalez N, Garcia S, Quintana JM. Factors related to functional prognosis in elderly patients after accidental hip fractures: a prospective cohort study. BMC Geriatr. 2014 Nov 26;14:124. doi: 10.1186/1471-2318-14-124. PMID 25425462
- [Background] Piscitelli P, Iolascon G, Argentiero A, Chitano G, Neglia C, Marcucci G, Pulimeno M, Benvenuto M, Mundi S, Marzo V, Donati D, Baggiani A, Migliore A, Granata M, Gimigliano F, Di Blasio R, Gimigliano A, Renzulli L, Brandi ML, Distante A, Gimigliano R. Incidence and costs of hip fractures vs strokes and acute myocardial infarction in Italy: comparative analysis based on national hospitalization records. Clin Interv Aging. 2012;7:575-83. doi: 10.2147/CIA.S36828. Epub 2012 Dec 17. PMID 23269863
- [Background] Marottoli RA, Berkman LF, Leo-Summers L, Cooney LM Jr. Predictors of mortality and institutionalization after hip fracture: the New Haven EPESE cohort. Established Populations for Epidemiologic Studies of the Elderly. Am J Public Health. 1994 Nov;84(11):1807-12. doi: 10.2105/ajph.84.11.1807. PMID 7977922
- [Background] French DD, Bass E, Bradham DD, Campbell RR, Rubenstein LZ. Rehospitalization after hip fracture: predictors and prognosis from a national veterans study. J Am Geriatr Soc. 2008 Apr;56(4):705-10. doi: 10.1111/j.1532-5415.2007.01479.x. Epub 2007 Nov 15. PMID 18005354
- [Background] Taylor BC, Schreiner PJ, Stone KL, Fink HA, Cummings SR, Nevitt MC, Bowman PJ, Ensrud KE. Long-term prediction of incident hip fracture risk in elderly white women: study of osteoporotic fractures. J Am Geriatr Soc. 2004 Sep;52(9):1479-86. doi: 10.1111/j.1532-5415.2004.52410.x. PMID 15341549
- [Background] Davenport SJ, Arnold M, Hua C, Schenck A, Batten S, Taylor NF. Physical Activity Levels During Acute Inpatient Admission After Hip Fracture are Very Low. Physiother Res Int. 2015 Sep;20(3):174-81. doi: 10.1002/pri.1616. Epub 2014 Dec 4. PMID 25475700
- [Background] Tudor-Locke C, Burton NW, Brown WJ. Leisure-time physical activity and occupational sitting: Associations with steps/day and BMI in 54-59 year old Australian women. Prev Med. 2009 Jan;48(1):64-8. doi: 10.1016/j.ypmed.2008.10.016. Epub 2008 Oct 30. PMID 19027786
- [Background] Macera CA, Hootman JM, Sniezek JE. Major public health benefits of physical activity. Arthritis Rheum. 2003 Feb 15;49(1):122-8. doi: 10.1002/art.10907. No abstract available. PMID 12579603
- [Background] Roy MA, Doherty TJ. Reliability of hand-held dynamometry in assessment of knee extensor strength after hip fracture. Am J Phys Med Rehabil. 2004 Nov;83(11):813-8. doi: 10.1097/01.phm.0000143405.17932.78. PMID 15502733
- [Background] Leino KA, Kuusniemi KS, Lertola KK, Olkkola KT. Comparison of four pain scales in patients with hip fracture or other lower limb trauma. Acta Anaesthesiol Scand. 2011 Apr;55(4):495-502. doi: 10.1111/j.1399-6576.2010.02373.x. Epub 2011 Feb 2. PMID 21288225
- [Background] Hollman JH, Beckman BA, Brandt RA, Merriwether EN, Williams RT, Nordrum JT. Minimum detectable change in gait velocity during acute rehabilitation following hip fracture. J Geriatr Phys Ther. 2008;31(2):53-6. doi: 10.1519/00139143-200831020-00003. PMID 19856550
- [Result] Corna S, Arcolin I, Giardini M, Bellotti L, Godi M. Addition of aerobic training to conventional rehabilitation after hip fracture: a randomized, controlled, pilot feasibility study. Clin Rehabil. 2021 Apr;35(4):568-577. doi: 10.1177/0269215520968694. Epub 2020 Nov 1. PMID 33131328
- [Derived] Fairhall NJ, Dyer SM, Mak JC, Diong J, Kwok WS, Sherrington C. Interventions for improving mobility after hip fracture surgery in adults. Cochrane Database Syst Rev. 2022 Sep 7;9(9):CD001704. doi: 10.1002/14651858.CD001704.pub5. PMID 36070134